CLINICAL TRIAL: NCT05580718
Title: Online Cognitive Behavioral Therapy Targeting Cardiac Anxiety Following Myocardial Infarction: A Randomized Controlled Trial
Brief Title: Online Cognitive Behavioral Therapy Targeting Cardiac Anxiety
Acronym: MI-CBT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Swedish Heart Lung Foundation (Other); The Swedish Research Council (Other Government); Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Josefin Särnholm, Principal Investigator, PhD, Karolinska Institutet
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MI-RCT1
Record Dates: First submitted 2022-10-07; First posted 2022-10-14 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Online CBT Targeting Cardiac Anxiety
Keywords: Myocardial infarction; Cardiac Anxiety; internet-CBT; Secondary prevention
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online CBT targeting cardiac anxiety (Experimental): CBT for MI primarily targets two processes of MI-related disability: fear of cardiac-related symptoms avoidance behavior and physical inactivity. The CBT is therapist-guided and lasts for 8 weeks.
  Interventions: Behavioral: MI-CBT
- Waitlist control (No Intervention): Participants randomised to waitlist can have no other concurrent psychological treatment but are free to use any medical treatment as usual. Participants on the waitlist also complete pre- and post-treatment, the follow-up measurement as well as weekly instruments (with exception of the treatment process measures Credibility scale and WAI). After the 3-month follow-up assessments, participants will receive internet-CBT for MI over 8 weeks

INTERVENTIONS:
Behavioral: MI-CBT — * Education Common reactions following MI and general lifestyle advice on e.g., physical activity. The role of cardiac anxiety and avoidance behavior on quality of life and physical health. Brief training in self-observation.
  * Goal setting Identifying life areas impaired by MI-related disability or symptom fear. Set health behavioral goals i.e., increased physical activity and gradually take steps towards them.
  * Exposure therapy Exposure to physical sensations (e.g., palpitations due to physical activity) to reduce fear of these symptoms. Gradual exposure to avoided situations, activities and increase in physical activity.
  * Relapse prevention Prevention of relapse into avoidance behaviors by identifying risk situations and conduct a plan forward on maintaining a healthy physically and active lifestyle.
  Arms: Online CBT targeting cardiac anxiety

SUMMARY:
The purpose of the present study is to evaluate an internet-delivered exposure-based cognitive behavioral therapy (CBT) protocol tailored for patients following myocardial infaction (MI) to increase Quality of Life (Qol) and physical activity by reducing cardiac anxiety.

DETAILED DESCRIPTION:
In the present research project, the investigators have tailored a CBT protocol to target the hypothesized mechanisms of how cardiac anxiety affects the clinical course of MI; by using exposure therapy to reduce fear, hypervigilance, and misinterpretations of cardiac symptoms to reduce MI-related avoidance and increasing physical activity.

Participants (estimated N=100) are randomized to internet-delivered CBT for 8 weeks or to a waitlist offered treatment as usual. Patients in the control arm will be crossed over to CBT treatment 3 months after the experimental group has completed treatment. Assessments will be conducted pre-treatment, post-treatment, 3 months (primary endpoint), 1-, 2 - and 5 years after treatment. These measurement points will also include the control group as it is crossed over to CBT after the 3-month follow-up

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:
* Myocardial infarction ≥ 6 months before assessment (type 1 STEMI/NSTEMI)
* Age 18-80 years;
* Clinically significant cardiac anxiety that leads to severe distress and/or interferes with daily life
* On adequate medical treatment(21); (E) Able to read and write in Swedish.

Exclusion Criteria:

* heart failure with severe systolic dysfunction (ejection fraction ≤ 35%)
* Significant valvular disease
* Planned coronary artery bypass surgery or percutaneous interventions
* Any medical restriction to physical exercise
* Severe medical illness
* Grade 3 hypertension (i.e., blood pressure ≥ 180 systolic and/or 110 diastolic)
* Severe psychiatric disorder or risk of suicide
* Alcohol dependency
* Ongoing psychological treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2025-03-14 (Estimated); Study Completion 2025-03-14 (Estimated)

PRIMARY OUTCOMES:
Seattle Angina Questionnaire | From baseline to 5 months
  A measure of coronary artery disease on five scales: physical limitation scale, anginal stability scale, anginal frequency scale, treatment satisfaction scale, and the disease. perception scale with a score ranging from 0 to 100. A higher score indicating a better quality of life.

SECONDARY OUTCOMES:
Seattle Angina Questionnaire | From baseline to 8 weeks
  A measure of coronary artery disease on five scales: physical limitation scale, anginal stability scale, anginal frequency scale, treatment satisfaction scale, and the disease perception scale. With a score ranging from 0 to 100. A higher score indicating a better quality of life.
Seattle Angina Questionnaire | Change over 8 measurement points measured from baseline and weekly for 8 weeks during treatment
  A measure of coronary artery disease on five scales: physical limitation scale, anginal stability scale, anginal frequency scale, treatment satisfaction scale, and the disease perception scale. With a score ranging from 0 to 100. A higher score indicating a better quality of life.
Seattle Angina Questionnaire | From baseline to 1 year and 2 months
  A measure of coronary artery disease on five scales: physical limitation scale, anginal stability scale, anginal frequency scale, treatment satisfaction scale, and the disease perception scale. With a score ranging from 0 to 100. A higher score indicating a better quality of life.
Seattle Angina Questionnaire | From baseline to 2 years and 2 months
  A measure of coronary artery disease on five scales: physical limitation scale, anginal stability scale, anginal frequency scale, treatment satisfaction scale, and the disease perception scale. With a score ranging from 0 to 100. A higher score indicating a better quality of life
Seattle Angina Questionnaire | From baseline to 5 years and 2 months
  A measure of coronary artery disease on five scales: physical limitation scale, anginal stability scale, anginal frequency scale, treatment satisfaction scale, and the disease perception scale. With a score ranging from 0 to 100. A higher score indicating a better quality of life.
12-Item Short-Form Health Survey | From baseline to 8 weeks
  General quality of life, with a score ranging from 0 to 100. A higher score indicating a better quality of life
12-Item Short-Form Health Survey | From baseline to 5 months
  General quality of life, with a score ranging from 0 to 100. A higher score indicating a better quality of life
12-Item Short-Form Health Survey | From baseline to 1 year and 2 months
  General quality of life, with a score ranging from 0 to 100. A higher score indicating a better quality of life
12-Item Short-Form Health Survey | From baseline to 2 year and 2 months
  General quality of life, with a score ranging from 0 to 100. A higher score indicating a better quality of life
12-Item Short-Form Health Survey | From baseline to 5 year and 2 months
  General quality of life, with a score ranging from 0 to 100. A higher score indicating a better quality of life
Cardiac anxiety questionnaire | From baseline to 8 weeks
  Measure of cardiac anxiety, fear, avoidance and attention. The score ranges between 0 and 72, with a greater score indicating elevated cardiac anxiety.
Cardiac anxiety questionnaire | Change over 8 measurement points measured from baseline and weekly for 8 weeks during treatment
  Measure of cardiac anxiety, fear, avoidance and attention. The score ranges between 0 and 72, with a greater score indicating elevated cardiac anxiety.
Cardiac anxiety questionnaire | From baseline to 5 months
  Measure of cardiac anxiety, fear, avoidance and attention. The score ranges between 0 and 72, with a greater score indicating elevated cardiac anxiety.
Cardiac anxiety questionnaire | From baseline to 1 year and 2 months
  Measure of cardiac anxiety, fear, avoidance and attention. The score ranges between 0 and 72, with a greater score indicating elevated cardiac anxiety.
Cardiac anxiety questionnaire | From baseline to 2 year and 2 months
  Measure of cardiac anxiety, fear, avoidance and attention. The score ranges between 0 and 72, with a greater score indicating elevated cardiac anxiety.
Cardiac anxiety questionnaire | From baseline to 5 year and 2 months
  Measure of cardiac anxiety, fear, avoidance and attention. The score ranges between 0 and 72, with a greater score indicating elevated cardiac anxiety.
Myocardial infarction behavior questionnaire | From baseline to 8 weeks
  MI-related avoidance questionnaire behaviors developed by the research group
Myocardial infarction behavior questionnaire | From baseline to 5 months
  MI-related avoidance questionnaire behaviors developed by the research group
Myocardial infarction behavior questionnaire | From baseline to 1 year and 2 months
  MI-related avoidance questionnaire behaviors developed by the research group. score ranging from 0 to 68 . Higher scores indicate more avoidance behavior.
Myocardial infarction behavior questionnaire | From baseline to 2 years and 2 months
  MI-related avoidance questionnaire behaviors developed by the research group. score ranging from 0 to 68 . Higher scores indicate more avoidance behavior.
Myocardial infarction behavior questionnaire | From baseline to 5 years and 2 months
  MI-related avoidance questionnaire behaviors developed by the research group. score ranging from 0 to 68 . Higher scores indicate more avoidance behavior.
Body Sensation Questionnaire | From baseline to 8 weeks
  Fear of bodily symptoms, score ranging from 0 to 72 . Higher scores indicate more fear of body sensations.
Body Sensation Questionnaire | From baseline to 5 months
  Fear of bodily symptoms, score ranging from 0 to 72 . Higher scores indicate more fear of body sensations.
Body Sensation Questionnaire | From baseline to 1 year and 2 months
  Fear of bodily symptoms, score ranging from 0 to 72 . Higher scores indicate more fear of body sensations.
Body Sensation Questionnaire | From baseline to 2 years and 2 months
  Fear of bodily symptoms, score ranging from 0 to 72 . Higher scores indicate more fear of body sensations.
Body Sensation Questionnaire | From baseline to 5 years and 2 months
  Fear of bodily symptoms, score ranging from 0 to 72 . Higher scores indicate more fear of body sensations.
Symptom checklist Severity and Frequency Scale (SCL, adapted to coronary artery disease) | From baseline to 8 weeks
  Cardiac-related symptoms in two sub scales A) frequency: score ranging from 0-48, with higher score indicating higher frequency of symptoms, B) severity of experienced symptom: score ranging from 0- 48, with a higher score indicating more severe symptoms
Symptom checklist Severity and Frequency Scale (SCL, adapted to coronary artery disease) | From baseline to 5 months
  Cardiac-related symptoms in two sub scales A) frequency: score ranging from 0-48, with higher score indicating higher frequency of symptoms, B) severity of experienced symptom: score ranging from 0- 48, with a higher score indicating more severe symptoms
Symptom checklist Severity and Frequency Scale (SCL, adapted to coronary artery disease) | From baseline to 1 year and 2 months
  Cardiac-related symptoms in two sub scales A) frequency: score ranging from 0-48, with higher score indicating higher frequency of symptoms, B) severity of experienced symptom: score ranging from 0- 48, with a higher score indicating more severe symptoms
Symptom checklist Severity and Frequency Scale (SCL, adapted to coronary artery disease) | From baseline to 2 years and 2 months
  Cardiac-related symptoms in two sub scales A) frequency: score ranging from 0-48, with higher score indicating higher frequency of symptoms, B) severity of experienced symptom: score ranging from 0- 48, with a higher score indicating more severe symptoms
Symptom checklist Severity and Frequency Scale (SCL, adapted to coronary artery disease) | From baseline to 5 years and 2 months
  Cardiac-related symptoms in two sub scales A) frequency: score ranging from 0-48, with higher score indicating higher frequency of symptoms, B) severity of experienced symptom: score ranging from 0- 48, with a higher score indicating more severe symptoms
Patient Health Questionnaire-9 | From Baseline to 8 weeks
  Measure of depression, score ranging 0 to 27 with a higher score indicating higher level of depression
Patient Health Questionnaire-9 | From Baseline to 5 months
  Measure of depression, score ranging 0 to 27 with a higher score indicating higher level of depression
Patient Health Questionnaire-9 | From Baseline to 1 year and 2 months
  Measure of depression, score ranging 0 to 27 with a higher score indicating higher level of depression
Patient Health Questionnaire-9 | From Baseline to 2 years and 2 months
  Measure of depression, score ranging 0 to 27 with a higher score indicating higher level of depression
Patient Health Questionnaire-9 | From Baseline to 5 years and 2 months
  Measure of depression, score ranging 0 to 27 with a higher score indicating higher level of depression
Generalized Anxiety Disorder 7-item | From Baseline to 8 weeks
  General anxiety, score ranging from 0-21, with a higher score indicating more anxiety and worry.
Generalized Anxiety Disorder 7-item | From Baseline to 5 months
  General anxiety, score ranging from 0-21, with a higher score indicating more anxiety and worry.
Generalized Anxiety Disorder 7-item | From Baseline to 1 year and 2 months
  General anxiety, score ranging from 0-21, with a higher score indicating more anxiety and worry.
Generalized Anxiety Disorder 7-item | From Baseline to 2 years and 2 months
  General anxiety, score ranging from 0-21, with a higher score indicating more anxiety and worry.
Generalized Anxiety Disorder 7-item | From Baseline to 5 years and 2 months
  General anxiety, score ranging from 0-21, with a higher score indicating more anxiety and worry.
Perceived stress scale 4-item | Baseline to 8 weeks
  Stress reactivity. A greater score indicate more perceived stress.
Perceived stress scale 4-item | Baseline to 5 months
  Stress reactivity. Score ranges 0-16 and a greater score indicate more perceived stress.
Perceived stress scale 4-item | Baseline to 1 year and 2 months
  Stress reactivity. Score ranges 0-16 and a greater score indicate more perceived stress.
Perceived stress scale 4-item | Baseline to 2 years and 2 months
  Stress reactivity. Score ranges 0-16 and a greater score indicate more perceived stress.
Perceived stress scale 4-item | Baseline to 5 years and 2 months
  Stress reactivity. Score ranges 0-16 and a greater score indicate more perceived stress.
The Godin Leisure-time Exercise and International Physical Activity Questionnaire 1 item on inactivity | Baseline to 8 weeks
  Level of physical activity and inactivity: On the Godin leisure-time excercise: The participant rate numbers of time per week that they engage in physical activity. The numb ers are the categorized in to low, moderate, and high levels of physical activity. And from International Physical Activity Questionnaire we will use 1 item on inactivity
The Godin Leisure-time Exercise and International Physical Activity Questionnaire 1 item on inactivity | Baseline to 5 months
  Level of physical activity and inactivity: On the Godin leisure-time excercise: The participant rate numbers of time per week that they engage in physical activity. The numb ers are the categorized in to low, moderate, and high levels of physical activity. And from International Physical Activity Questionnaire we will use 1 item on inactivity
The Godin Leisure-time Exercise and International Physical Activity Questionnaire 1 item on inactivity | Baseline to 1 year and 2 months
  Level of physical activity and inactivity: On the Godin leisure-time excercise: The participant rate numbers of time per week that they engage in physical activity. The numb ers are the categorized in to low, moderate, and high levels of physical activity. And from International Physical Activity Questionnaire we will use 1 item on inactivity
The Godin Leisure-time Exercise and International Physical Activity Questionnaire 1 item on inactivity | Baseline to 2 years and 2 months
  Level of physical activity and inactivity: On the Godin leisure-time excercise: The participant rate numbers of time per week that they engage in physical activity. The numb ers are the categorized in to low, moderate, and high levels of physical activity. And from International Physical Activity Questionnaire we will use 1 item on inactivity
The Godin Leisure-time Exercise and International Physical Activity Questionnaire 1 item on inactivity | Baseline to 5 years and 2 months
  Level of physical activity and inactivity: On the Godin leisure-time excercise: The participant rate numbers of time per week that they engage in physical activity. The numb ers are the categorized in to low, moderate, and high levels of physical activity. And from International Physical Activity Questionnaire we will use 1 item on inactivity
Lifestyle factors: The national Board of health and Welfare questionnaire | Baseline to 8 weeks
  Questionnaire regarding diet (5 item), tobacco (2 item) and alcohol (3 item) diet (5 item), tobacco (2 item) and alcohol (3 item) and BMI.
Lifestyle factors: The national Board of health and Welfare questionnaire | Baseline to 5 months
  Questionnaire regarding diet (5 item), tobacco (2 item) and alcohol (3 item) diet (5 item), tobacco (2 item) and alcohol (3 item) and BMI.
Lifestyle factors: The national Board of health and Welfare questionnaire | Baseline to 1 year and 2 months
  Questionnaire regarding diet (5 item), tobacco (2 item) and alcohol (3 item) diet (5 item), tobacco (2 item) and alcohol (3 item) and BMI.
Lifestyle factors: The national Board of health and Welfare questionnaire | Baseline to 2 years and 2 months
  Questionnaire regarding diet (5 item), tobacco (2 item) and alcohol (3 item) diet (5 item), tobacco (2 item) and alcohol (3 item) and BMI.
Lifestyle factors: The national Board of health and Welfare questionnaire | Baseline to 5 years and 2 months
  Questionnaire regarding diet (5 item), tobacco (2 item) and alcohol (3 item) diet (5 item), tobacco (2 item) and alcohol (3 item) and BMI.
Healthcare consumption and work loss:Tic-P | From baseline to 8 weeks
  The Trimbos and Institute of Medical Technology Assessment Cost Questionnaire for Psychiatry assesses societal cost during the last month. These costs include the participant's health care consumption (direct medical costs), time spent in other health promoting activities (direct non-medical costs), and sick leave, unemployment, and reduced work capacity at work and in the domestic realm (indirect non-medical costs).
Healthcare consumption and work loss:Tic-P | From baseline to 5 months
  The Trimbos and Institute of Medical Technology Assessment Cost Questionnaire for Psychiatry assesses societal cost during the last month. These costs include the participant's health care consumption (direct medical costs), time spent in other health promoting activities (direct non-medical costs), and sick leave, unemployment, and reduced work capacity at work and in the domestic realm (indirect non-medical costs).
Healthcare consumption and work loss:Tic-P | From baseline to 1 year and 2 months
  The Trimbos and Institute of Medical Technology Assessment Cost Questionnaire for Psychiatry assesses societal cost during the last month. These costs include the participant's health care consumption (direct medical costs), time spent in other health promoting activities (direct non-medical costs), and sick leave, unemployment, and reduced work capacity at work and in the domestic realm (indirect non-medical costs).
Healthcare consumption and work loss:Tic-P | From baseline to 2 years and 2 months
  The Trimbos and Institute of Medical Technology Assessment Cost Questionnaire for Psychiatry assesses societal cost during the last month. These costs include the participant's health care consumption (direct medical costs), time spent in other health promoting activities (direct non-medical costs), and sick leave, unemployment, and reduced work capacity at work and in the domestic realm (indirect non-medical costs).
Healthcare consumption and work loss:Tic-P | From baseline to 5 years and 2 months
  The Trimbos and Institute of Medical Technology Assessment Cost Questionnaire for Psychiatry assesses societal cost during the last month. These costs include the participant's health care consumption (direct medical costs), time spent in other health promoting activities (direct non-medical costs), and sick leave, unemployment, and reduced work capacity at work and in the domestic realm (indirect non-medical costs).
University of Toronto Atrial fibrillation Severity Scale (AFSS) | From Baseline to 8 weeks
  3 item on cardiac-specific healthcare consumption. Scores ranges 0-15 with a higher score indicating more cardiac-related healthcare consumption.
University of Toronto Atrial fibrillation Severity Scale (AFSS) | From Baseline to 5 months
  3 item on cardiac-specific healthcare consumption. Scores ranges 0-15 with a higher score indicating more cardiac-related healthcare consumption.
University of Toronto Atrial fibrillation Severity Scale (AFSS) | From Baseline to 1 year and 2 months
  3 item on cardiac-specific healthcare consumption. Scores ranges 0-15 with a higher score indicating more cardiac-related healthcare consumption.
University of Toronto Atrial fibrillation Severity Scale (AFSS) | From Baseline to 2 years and 2 months
  3 item on cardiac-specific healthcare consumption. Scores ranges 0-15 with a higher score indicating more cardiac-related healthcare consumption.
University of Toronto Atrial fibrillation Severity Scale (AFSS) | From Baseline to 5 years and 2 months
  3 item on cardiac-specific healthcare consumption. Scores ranges 0-15 with a higher score indicating more cardiac-related healthcare consumption.

OTHER OUTCOMES:
Number of Participants With Abnormal Laboratory Values | From Baseline to 8 weeks
  Venous blood will be collected for local analyses of fasting plasma glucose, HbA1c, plasma total cholesterol, LDL, HDL, triglycerides, hsCRP, creatinine, stress-related hormones such as cortisol, copeptin and vasopressin
Number of Participants With Abnormal Laboratory Values | From Baseline to 5 months
  Venous blood will be collected for local analyses of fasting plasma glucose, HbA1c, plasma total cholesterol, LDL, HDL, triglycerides, hsCRP, creatinine, stress-related hormones such as cortisol, copeptin and vasopressin
Algometry (Somedic AB, Hörby, Sweden) | From Baseline to 8 weeks
  A pain sensitivity measurement with algometry (Somedic AB, Hörby, Sweden); consisting of a handle with a 1 cm rubber plate at the end will be used. Algometers are used to measure pressure pain thresholds, the exact pressure (kPa) is registered in the algometer and thus a measure of a person's pain threshold can be assessed.
Algometry (Somedic AB, Hörby, Sweden) | From Baseline to 5 months
  A pain sensitivity measurement with algometry (Somedic AB, Hörby, Sweden); consisting of a handle with a 1 cm rubber plate at the end will be used. Algometers are used to measure pressure pain thresholds, the exact pressure (kPa) is registered in the algometer and thus a measure of a person's pain threshold can be assessed.
Accelerometer (Actigraf®) | Baseline to 8 weeks
  An Accelerometer (Actigraf®) will be carried on the wrist over to measure physical activity over 1 week
Accelerometer (Actigraf®) | Baseline to 5 months
  An Accelerometer (Actigraf®) will be carried on the wrist over to measure physical activity over 1 week week at each assessment
Adverse events | From Baseline to 8 weeks
  Potential adverse reactions to the treatment. Participants will be asked to report and rate the short- and long term discomfort of the adverse event on a scale from 0 ('did not affect me at all') and 3 ('affected me very negatively').
Adverse events | 8 measurement points measured from baseline and weekly for 8 weeks during treatment
  Potential adverse reactions to the treatment. Participants will be asked to report and rate the short- and long term discomfort of the adverse event on a scale from 0 ('did not affect me at all') and 3 ('affected me very negatively').
Adverse events | From Baseline to 5 months
  Potential adverse reactions to the treatment. Participants will be asked to report and rate the short- and long term discomfort of the adverse event on a scale from 0 ('did not affect me at all') and 3 ('affected me very negatively').
Adverse events | From Baseline to 1 year and 2 months
  Potential adverse reactions to the treatment. Participants will be asked to report and rate the short- and long term discomfort of the adverse event on a scale from 0 ('did not affect me at all') and 3 ('affected me very negatively').
Adverse events | From Baseline to 2 years and 2 months
  Potential adverse reactions to the treatment. Participants will be asked to report and rate the short- and long term discomfort of the adverse event on a scale from 0 ('did not affect me at all') and 3 ('affected me very negatively').
Adverse events | From Baseline to 5 years and 2 months
  Potential adverse reactions to the treatment. Participants will be asked to report and rate the short- and long term discomfort of the adverse event on a scale from 0 ('did not affect me at all') and 3 ('affected me very negatively').
Client satisfaction Questionnaire | Baseline to 8 weeks
  Treatment satisfaction, score ranging from 0 to 32, with a higher score indication more satisfaction with the treatment.
Treatment Credibility Scale | 1-2 weeks from baseline
  Measures treatment credibility
Working Alliance Inventory | 1-2 weeks from baseline
  Measures therapeutic alliance with the psychologist
Follow-up questions on health changes | Baseline to 8 weeks
  We will ask participant to describe if they have experienced any psychosocial stressors, changes in physical health, such as invasive therapy and changes of medication
Follow-up questions on health changes | Baseline to 5 months
  We will ask participant to describe if they have experienced any psychosocial stressors, changes in physical health, such as invasive therapy and changes of medication
Follow-up questions on health changes | Baseline to 1 year and 2 months
  We will ask participant to describe if they have experienced any psychosocial stressors, changes in physical health, such as invasive therapy and changes of medication
Follow-up questions on health changes | Baseline to 2 years and 2 months
  We will ask participant to describe if they have experienced any psychosocial stressors, changes in physical health, such as invasive therapy and changes of medication
Follow-up questions on health changes | Baseline to 5 years and 2 months
  We will ask participant to describe if they have experienced any psychosocial stressors, changes in physical health, such as invasive therapy and changes of medication
AFFS/SCL-4 | Change over 8 measurement points measured from baseline and weekly for 8 weeks during treatment
  4 items derived from the Symptoms Checklist (SCL) and the Atrial Fibrillation Severity Scale (AFSS) measuring disabling cardiac symptoms
MI-behavior Questionnaire | Change over 8 measurement points measured from baseline and weekly for 8 weeks during treatment
  5 items measuring avoidance behavior from the MI-related avoidance questionnaire behaviors developed by the research group
Perceived stress scale 4-item | Change over 8 measurement points measured from baseline and weekly for 8 weeks during treatment
  Measure of perceived stress and stress reactivity. Score ranging 0 -16 with a higher score indicating more perceived stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-06-18): https://cdn.clinicaltrials.gov/large-docs/18/NCT05580718/SAP_000.pdf